CLINICAL TRIAL: NCT03005990
Title: The Effects of Exercise Training in Community-dwelling Elderly With Sleep Disturbances With Follow-up: Body Composition and Energy Metabolism
Brief Title: The Effects of Exercise Training in Community-dwelling Elderly With Sleep Disturbances With Follow-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201512210RIND
Record Dates: First submitted 2016-12-13; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Exercise Addiction; Sleep Disorder
Keywords: Sleep disturbance; Body composition; Energy metabolism; Exercise training; Community-dwelling elderly
MeSH Terms: conditions — Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training group (Experimental): Exercise group will attend a supervised aerobic plus resistance exercise training class 3 times a week totally for 24 weeks.
  Interventions: Other: Exercise training group
- Control group (No Intervention): Control group only provide standard outpatient care program.

INTERVENTIONS:
Other: Exercise training group — The conditioning period (24 weeks) of the exercise intervention was under the supervision of an exercise physiologist. The conditioning protocol included aerobic exercise sessions 3 times per week with 70-85% of maximal heart rate(max HR) for 30 mins and resistance sessions 3 times per week with an intensity of 80% of one-repetition maximum(1RM), 3 sets of 8 repetitions maximum. Each participant will measured the borg rating of perceived exertion scale and heart rate monitor during exercise. Exercise sessions were conducted in the afternoon (3-5 PM).
  Arms: Exercise training group

SUMMARY:
This study will explore the long-term effects of exercise training on body composition, cardiorespiratory fitness, and energy metabolism in the community-dwelling elderly with sleep disturbances

DETAILED DESCRIPTION:
This project will be conducted in three years:

In the first year,investigators will explore the correlation of sleep parameters, dietary behavior and body composition in community-dwelling elders. Two hundred elders will be recruited to receive the actigraph accelerometer recording, sleep quality questionnaire, bio-electrical impedance analysis, heart rate variability analysis, cognitive and depression evaluation.

Secondly, the study will evaluate the efficacy and possible mechanisms of a 24-week exercise training for sleep disturbances patients. Sixty patients with sleep disturbances elders will be randomized to exercise group or control group. Participants in the exercise group will receive aerobic and resistance exercise 3 times per week for 24 weeks. The controls will receive sleep hygiene education and consultation. All measurements will be performed as described before.

Finally, all the 260 elders participating in this study will receive 12-month follow-up assessments to explore the longitudinal impact of sleep disturbances on cardiorespiratory function, body composition and metabolic function, and long-term effect of exercise training on sleep disturbances patients. Investigators expect elders with poor sleep quality have lower level of health-related fitness and metabolic function; exercise training is effective to improve sleep quality, metabolic function and general health in the elders with sleep disturbances, and the effect can be sustained for a long period.

ELIGIBILITY:
Inclusion Criteria:

1. Community dwelling sedentary men and women who were 65 years or older

Exclusion Criteria:

1. History of Diagnostic and Statistical Manual Diploma in Social Medicine, 4th. Edition (DSM-IV) criteria for any major psychiatric disorder, including mania or alcohol or substance abuse
2. History of cognitive or other neurological disorders
3. Other sleep disorders by history or documented on screening polysomnography (apnea index >10, periodic leg movement arousal index >15, or rapid eye movement (REM) behavior disorder
4. Unstable or serious medical conditions or cardiopulmonary disease that contraindicate exercise
5. BMI > 35 kg/m2
6. Individual with a life expectancy of no more than 1 years or final stage of cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Body fat percentage | Up to 1 year (the first year)
  Body fat percentage in percentage.

SECONDARY OUTCOMES:
Body fat mass | Up to 1 year (the first year)
  Body fat mass in kilograms.
Body fat free mass | Up to 1 year (the first year)
  Body fat free mass in kilograms.
Body mass index | Up to 1 year (the first year)
  BMI in kg/m^2.
Rest metabolic rate | Up to 1 year (the first year)
  Rest metabolic rate in percentage.
Impedance | Up to 1 year (the first year)
  Impedance in ohm.
Resistance | Up to 1 year (the first year)
  Resistance in ohm.
Electroencephalography(EEG) | Pretest and after 24 weeks intervention (the second year)
  Electroencephalography was assessed during sleep.
Electrooculography(EOG) | Pretest and after 24 weeks intervention (the second year)
  Electrooculography was assessed during sleep.
Electromyography(EMG) | Pretest and after 24 weeks intervention (the second year)
  Electromyography was assessed during sleep.
Electrocardiography(ECG) | Pretest and after 24 weeks intervention (the second year)
  Electrocardiography was assessed during sleep.
Pittsburgh sleep quality index | Up to 1 year (the first year)
Dual energy X-ray absorptiometry | Pretest and after 24 weeks intervention (the second year)
Triglyceride | Pretest and after 24 weeks intervention (the second year)
  Triglyceride in mg/dL.
Total cholesterol | Pretest and after 24 weeks intervention (the second year)
  Total cholesterol in mg/dL.
Insulin | Pretest and after 24 weeks intervention (the second year)
  Insulin in uIU/mL.
Fasting glucose | Pretest and after 24 weeks intervention (the second year)
  Fasting glucose in mg/dL.
Glycated hemoglobin(HbA1C) | Pretest and after 24 weeks intervention (the second year)
  HbA1C in percentage.
High-density lipoprotein | Pretest and after 24 weeks intervention (the second year)
  High-density lipoprotein in mg/dL.
Low-density lipoprotein | Pretest and after 24 weeks intervention (the second year)
  Low-density lipoprotein in mg/dL.
C-reactive protein | Pretest and after 24 weeks intervention (the second year)
  C-reactive protein in mg/dL.
Heart rate variability | Pretest and after 24 weeks intervention (the second year)
  It is measured by the variation in the beat-to-beat interval. Methods used to detect beats is electrocardiography.
Maximum oxygen consumption | Pretest and after 24 weeks intervention (the second year)
  Use treadmill exercise testing.
Three factor eating questionnaire | Up to 1 year (the first year)
Taiwan Geriatric Depression Scale | Up to 1 year (the first year)
Groningen Activity Restriction Scale | Up to 1 year (the first year)

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, doctor, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tseng TH, Chen HC, Wang LY, Chien MY. Effects of exercise training on sleep quality and heart rate variability in middle-aged and older adults with poor sleep quality: a randomized controlled trial. J Clin Sleep Med. 2020 Sep 15;16(9):1483-1492. doi: 10.5664/jcsm.8560. PMID 32394890